CLINICAL TRIAL: NCT07307638
Title: A Randomized, Double-blind, Placebo-controlled, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of ZT006 as Well as the Food Effect on the Pharmacokinetics of ZT006 in Healthy, Overweight and Obese Participants
Brief Title: Dose-escalation and Food Effect Study of ZT006 in Healthy, Overweight and Obese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing QL Biopharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BJQL-ZT006-1001
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Overweight,Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- ZT006 tablet, dose level 1, single dose, fasted (Experimental)
  Interventions: Drug: ZT006
- ZT006 tablet, dose level 2, single dose, fasted (Experimental)
  Interventions: Drug: ZT006
- ZT006 tablet, dose level 3, single dose, fasted (Experimental)
  Interventions: Drug: ZT006
- ZT006 tablet, dose level 4, single dose, fasted and fed (Experimental)
  Interventions: Drug: ZT006
- ZT006 tablet, dose level 5, single dose, fasted (Experimental)
  Interventions: Drug: ZT006
- ZT006 tablet, multiple doses, cohort 1 (Experimental)
  Interventions: Drug: ZT006
- ZT006 tablet, multiple doses, cohort 2 (Experimental)
  Interventions: Drug: ZT006
- ZT006 tablet, multiple doses, cohort 3 (Experimental)
  Interventions: Drug: ZT006
- ZT006 tablet, multiple doses, cohort 4 (Experimental)
  Interventions: Drug: ZT006
- placebo of ZT006, single dose, fasted (Placebo Comparator)
  Interventions: Drug: Placebo of ZT006
- placebo of ZT006, single dose, fasted and fed (Placebo Comparator)
  Interventions: Drug: Placebo of ZT006
- placebo of ZT006, multiple doses (Placebo Comparator)
  Interventions: Drug: Placebo of ZT006

INTERVENTIONS:
Drug: ZT006 — Participants will receive a single dose of ZT006 of dose level 1 under fasted condition.
  Arms: ZT006 tablet, dose level 1, single dose, fasted
Drug: ZT006 — Participants will receive a single dose of ZT006 of dose level 2 under fasted condition.
  Arms: ZT006 tablet, dose level 2, single dose, fasted
Drug: ZT006 — Participants will receive a single dose of ZT006 of dose level 3 under fasted condition.
  Arms: ZT006 tablet, dose level 3, single dose, fasted
Drug: ZT006 — Participants will receive a single dose of ZT006 of dose level 4 under fasted condition in period 1, and after a high fat, high caloric breakfast in period 2.
  Arms: ZT006 tablet, dose level 4, single dose, fasted and fed
Drug: ZT006 — Participants will receive a single dose of ZT006 of dose level 5 under fasted condition.
  Arms: ZT006 tablet, dose level 5, single dose, fasted
Drug: ZT006 — Participants will receive daily doses of ZT006 for 42 days: dose level 1 for 7 days, then dose level 2 for 7 days, then dose level 3 for 28 days.
  Arms: ZT006 tablet, multiple doses, cohort 1
Drug: ZT006 — Participants will receive daily doses of ZT006 for 42 days: dose level 1 for 7 days, then dose level 2 for 7 days, then dose level 3 for 14 days, then dose level 4 for 14 days.
  Arms: ZT006 tablet, multiple doses, cohort 2
Drug: ZT006 — Participants will receive daily doses of ZT006 for 42 days: dose level 2 for 7 days, then dose level 3 for 7 days, then dose level 4 for 28 days.
  Arms: ZT006 tablet, multiple doses, cohort 3
Drug: ZT006 — Participants will receive daily doses of ZT006 for 42 days: dose level 2 for 7 days, then dose level 3 for 7 days, then dose level 4 for 14 days, then dose level 5 for 14 days.
  Arms: ZT006 tablet, multiple doses, cohort 4
Drug: Placebo of ZT006 — Participants will receive a single dose of placebo of ZT006 under fasted condition.
  Arms: placebo of ZT006, single dose, fasted
Drug: Placebo of ZT006 — Participants will receive a single dose of placebo of ZT006 under fasted condition in period 1, and after a high fat, high caloric breakfast in period 2.
  Arms: placebo of ZT006, single dose, fasted and fed
Drug: Placebo of ZT006 — Participants will receive daily doses of placebo of ZT006 for 42 days.
  Arms: placebo of ZT006, multiple doses

SUMMARY:
ZT006 is an oral, long-acting glucagon-like peptide-1. This first-in-human study is designed to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of ZT006 in healthy, overweight and obese participants. The study comprises three parts, i.e. single dose-escalation, multiple dose-escalation, food effect on the pharmacokinetics of ZT006.

In the single dose-escalation study, participants will receive a single dose (ZT006 dose level 1 - 5 or corresponding placebo) of ZT006 under fasted condition. A higher dose can only be given after obtaining acceptable safety and tolerability data for at least 7 days after the previous dose. After study drug administration, there will be a 7-day in-house period for safety observation and pharmacokinetics samples collection. Participants will join ambulatory visits until 42 days post-dose.

In the multiple dose-escalation study, participants will receive a daily dose of ZT006 or corresponding placebo over 42 days in a dose up-titration fashion according to the following regimen:

* Cohort 1: dose level 1 - dose level 2 - dose level 3
* Cohort 2: dose level 1 - dose level 2 - dose level 3 - dose level 4
* Cohort 3: dose level 2 - dose level 3 - dose level 4
* Cohort 4: dose level 2 - dose level 3 - dose level 4 - dose level 5

Dosing of a cohort with higher drug exposure can only be done after evaluation of safety and tolerability data for at least 14 days after the first dose in the previous cohort. Participants will join ambulatory visits until 35 days after the last dose.

To evaluate the food effect on the pharmacokinetics of ZT006, participants who have received single dose of ZT006 or placebo of dose level 4 in the single dose-escalation study will receive another dose of ZT006 or placebo after a high fat, high caloric breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, 12-lead electrocardiogram and clinical laboratory tests (hematology, urinalysis, chemistry, coagulation), as judged by the investigator.
* Male or female, age between 18 - 55 years (both inclusive) at the time of signing of the informed consent.
* Body mass index (BMI) 19.0 - 35.0 kg/m²(both inclusive). Body weight >50.0 kg for male participants and >45.0 kg for female participants. BMI 19 - 28.0 kg/m²(both inclusive) for single-dose escalation study, BMI 19.0 - 28.0 kg/m²(both inclusive) for cohorts 1 and 2 of multiple-dose escalation study, BMI 24.0 - 35.0 kg/m²(both inclusive) for cohorts 3 and 4 of multiple-dose escalation study.
* Having dietary caloric restriction and increased physical activity for ≥3 months, with change in body weight (increase or decrease) no more than 5%, irrespective of medical records.

Exclusion Criteria:

* Known hypersensitivity to the study drug or excipients or GLP-1 receptor agonists.
* Medical history of hypoglycemia.
* History or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2, or history of pancreatitis or symptomatic gallbladder disease.
* Previous diagnosis of endocrine disorders or monogenic mutations causing obesity, including but not limited to hypothalamic obesity, pituitary obesity, hypothyroidism-induced obesity, Cushing's syndrome, insulinoma, acromegaly, or hypogonadism.
* Use of GLP-1 receptor agonists within 30 days or 5 half-lives (whichever is longer) before the first dose of the investigational intervention.
* Glycated hemoglobin (HbA1c) > 6.0% or fasting plasma glucose < 3.9 mmol/L or > 6.1 mmol/L at screening, or diagnosed with diabetes mellitus of type 1 or type 2 diabetes or other specific types derived from other causes.
* Aspartate aminotransferase ≥ 2 × upper limit of normal (ULN), Alanine aminotransferase ≥ 2 × ULN, or total bilirubin ≥ 1.5 × ULN
* Calcitonin above ULN at screening.
* Other clinically significant diseases detected within 12 months before screening (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, pulmonary, immunological, psychiatric, or cardiovascular diseases).
* Use of prescription drugs (excluding topical eye/nose drops and creams without systemic exposure risk), over-the-counter drugs, dietary supplements, vitamins, or herbal medicines (excluding routine vitamins) within 2 weeks before screening.
* Long-term use of medications directly affecting gastrointestinal motility prior to screening. Use of weight-loss medications (including but not limited to orlistat) within 3 months before dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-06-14 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Rate of treatment-emergent adverse events after single dose administration under fasted condition. | From baseline to Day 43
  Summarized from adverse event reporting in %
Rate of treatment-emergent adverse events during and after multiple-dose administration. | From baseline to end of study (Day 77)
  Summarized from adverse event reporting in %
Rate of treatment-emergent adverse events after single dose administration under fed condition. | From Day 44 to end of study (Day 86)
  Summarized from adverse event reporting in %

SECONDARY OUTCOMES:
Area under the concentration-time curve from time zero to infinity after single-dose administration under fasted condition. | From baseline to Day 43
  Measured in ng*h/mL
Maximal observed concentration after single-dose administration under fasted condition. | From baseline to Day 43
  Measured in ng/mL
Time to reach the maximal observed concentration after single-dose administration under fasted condition. | From baseline to Day 43
  Measured in hours
Terminal half-life after single-dose administration under fasted condition. | From baseline to Day 43
  Measured in hours
Area under the concentration-time curve during the dosing interval at steady state. | Day 42 to Day 77
  Measured in ng*h/mL
Maximal observed concentration at steady state. | Day 42 to Day 77
  Measured in ng/mL
Time to reach the maximal observed concentration at steady state. | From Day 42 to Day 77
  Measured in hours
Terminal half-life at steady state. | From Day 42 to Day 77
  Measured in hours
Area under the concentration-time curve from time zero to infinity after single-dose administration under fed condition. | From Day 44 to end of study (Day 86)
  Measured in ng*h/mL
Maximal observed concentration after single-dose administration under fed condition. | From Day 44 to end of study (Day 86)
  Measured in ng/mL
Time to reach the maximal observed concentration after single-dose administration under fed condition. | From Day 44 to end of study (Day 86)
  Measured in hours
Terminal half-life after single-dose administration under fed condition. | From Day 44 to end of study (Day 86)
  Measured in hours
Incidence of ZT006 anti-drug antibody after single-dose administration under fasted condition. | From baseline to Day 43
  Measured in %
Incidence of ZT006 anti-drug antibody during and after multiple-dose administration. | From baseline to end of study (Day 77)
  Measured in %

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hu, MD, Principal Investigator — The Second Hospital of Anhui Medical University; Yijun Du, Master, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China